CLINICAL TRIAL: NCT06363643
Title: Lower Limb Arthroplasty: Effects of a Tele Prehabilitation Program With Indirect Electrostimulation. Randomized Controlled Clinical Trial
Brief Title: Lower Limb Arthroplasty: Effects of a Tele Prehabilitation Program With Indirect Electrostimulation.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Prehab01
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Osteo Arthritis Knee and Hip; Lower Limb Arthroplasty
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ELECTROSTIMULATION (ESM) (Experimental): ESM will perform the Tele Prehab program based on indirect electrostimulation.
  Interventions: Device: ELECTROSTIMULATION (ES)
- EXERCISE (C) (Active Comparator): Group C will perform the Tele Prehab program based on supervised exercise.
  Interventions: Other: EXERCISE (C)

INTERVENTIONS:
Device: ELECTROSTIMULATION (ES) — ES will receive the electrostimulator directly at home and will do three weekly Tele supervised sessions of 30 minutes of indirect electrostimulation. The treatment will last 4 weeks.
  Arms: ELECTROSTIMULATION (ESM)
Other: EXERCISE (C) — C will perform three weekly Tele supervised sessions of exercise. The treatment will last 4 weeks.
  Arms: EXERCISE (C)

SUMMARY:
Preoperative fitness is known to predict postoperative outcomes following lower limb arthroplasty, but many patients, especially the most fragile, arrive at surgery with reduced mobility and functional capacity.

Prehabilitation (Prehab) encompasses a series of interventions that are intended to help patients improve their physical state and psychological well-being pre-intervention to reduce the days of hospitalization and the number of post-operative complications. Patients who participate in Prehab require less postoperative care and consequently have less impact on the cost of the healthcare system. However, adherence to a face-to-face program is usually poor and presents both organizational and psychophysical barriers. In the last years, telerehabilitation has proven to be a viable alternative to face-to-face treatment and has already been adopted for the Prehab. Electrostimulation (ESM) is regularly used successfully in clinical settings for the recovery of muscle tone in patients with orthopedic pathologies. In addition, it has already been used for Prehab, showing an increase in muscle strength and a decrease in postoperative hospital stay following knee arthroplasty. Also Exercise offers benefits in the treatment of orthopedic patients because improve: strength, cardiovascular fitness, functional capacities and quality of life. Therefore, in a group of patients who are candidates for elective lower limb arthroplasty surgery, it was decided to evaluate the effects of a Tele Prehab program, based on the ESM, and compare them with those of an Tele Prehab exercise program, equal in dose and duration. The proposal differs from those present in the literature for complete administration in telerehabilitation, including evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Elective Knee or Total Hip arthroplasty

Exclusion Criteria:

* concomitant orthopaedic or neurological pathologies (other than the pathology for which arthroplasty has been indicated) that modify the ability to walk;
* pathologies that modify the balance (neurological and/or vestibular);
* contraindications to the use of medical equipment used in the study;
* inability to understand and sign informed consent.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-04-22 (Estimated); Primary Completion 2024-07-26 (Estimated); Study Completion 2024-07-26 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in functional capacities on 30 Seconds Chair Stand Test (30CST) at week 4 | Baseline and week 4
  30CST is a validated tool to assess strength and endurance of Lower limbs. The patient is seated in a 17" high chair. Count the number of times the patient comes to a full standing position in 30 seconds.

SECONDARY OUTCOMES:
Change from baseline in functional capacities on Timed Up and Go test (TUG) at week 4. | Baseline and week 4
  TUG is a validated tool to assess dynamic balance and functional mobility. The patient getting up from a chair from the sitting to the bipedal position, walking three meters, turning, returning, and sitting on the chair again. The variable measured is the total time, in seconds, taken by the test.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Marin, PhD, Principal Investigator — University of Pavia (Italy)
Locations (1):
- "Città di Pavia Healthcare Institute", Pavia, Italy

IPD SHARING:
Plan to Share IPD: Yes
The material will be shared as an attachment to the article. All the tools used in the study will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available when the article is published.
Access Criteria: Free access

REFERENCES:
- [Background] Bhave A, Marker DR, Seyler TM, Ulrich SD, Plate JF, Mont MA. Functional problems and treatment solutions after total hip arthroplasty. J Arthroplasty. 2007 Sep;22(6 Suppl 2):116-24. doi: 10.1016/j.arth.2007.04.025. Epub 2007 Jul 26. PMID 17823029
- [Background] Coudeyre E, Jardin C, Givron P, Ribinik P, Revel M, Rannou F. Could preoperative rehabilitation modify postoperative outcomes after total hip and knee arthroplasty? Elaboration of French clinical practice guidelines. Ann Readapt Med Phys. 2007 Apr;50(3):189-97. doi: 10.1016/j.annrmp.2007.02.002. Epub 2007 Feb 15. PMID 17343953
- [Background] Rooks DS, Huang J, Bierbaum BE, Bolus SA, Rubano J, Connolly CE, Alpert S, Iversen MD, Katz JN. Effect of preoperative exercise on measures of functional status in men and women undergoing total hip and knee arthroplasty. Arthritis Rheum. 2006 Oct 15;55(5):700-8. doi: 10.1002/art.22223. PMID 17013852
- [Background] Snow R, Granata J, Ruhil AV, Vogel K, McShane M, Wasielewski R. Associations between preoperative physical therapy and post-acute care utilization patterns and cost in total joint replacement. J Bone Joint Surg Am. 2014 Oct 1;96(19):e165. doi: 10.2106/JBJS.M.01285. PMID 25274793
- [Background] Desmeules F, Hall J, Woodhouse LJ. Prehabilitation improves physical function of individuals with severe disability from hip or knee osteoarthritis. Physiother Can. 2013 Spring;65(2):116-24. doi: 10.3138/ptc.2011-60. PMID 24403671
- [Background] Saw MM, Kruger-Jakins T, Edries N, Parker R. Significant improvements in pain after a six-week physiotherapist-led exercise and education intervention, in patients with osteoarthritis awaiting arthroplasty, in South Africa: a randomised controlled trial. BMC Musculoskelet Disord. 2016 May 27;17:236. doi: 10.1186/s12891-016-1088-6. PMID 27233479
- [Background] Karimijashni M, Yoo S, Barnes K, Poitras S. Pre- and Post-Operative Rehabilitation Interventions in Patients at Risk of Poor Outcomes Following Knee or Hip Arthroplasty: Protocol for Two Systematic Reviews. Adv Rehabil Sci Pract. 2023 May 10;12:27536351231170956. doi: 10.1177/27536351231170956. eCollection 2023 Jan-Dec. PMID 37188054
- [Background] De Klerk TC, Dounavi DM, Hamilton DF, Clement ND, Kaliarntas KT. Effects of home-based prehabilitation on pre- and postoperative outcomes following total hip and knee arthroplasty. Bone Jt Open. 2023 May 5;4(5):315-328. doi: 10.1302/2633-1462.45.BJO-2023-0021. PMID 37142259
- [Background] Walls RJ, McHugh G, O'Gorman DJ, Moyna NM, O'Byrne JM. Effects of preoperative neuromuscular electrical stimulation on quadriceps strength and functional recovery in total knee arthroplasty. A pilot study. BMC Musculoskelet Disord. 2010 Jun 14;11:119. doi: 10.1186/1471-2474-11-119. PMID 20540807
- [Background] Talbot LA, Gaines JM, Ling SM, Metter EJ. A home-based protocol of electrical muscle stimulation for quadriceps muscle strength in older adults with osteoarthritis of the knee. J Rheumatol. 2003 Jul;30(7):1571-8. PMID 12858461
- [Background] Lyons CL, Robb JB, Irrgang JJ, Fitzgerald GK. Differences in quadriceps femoris muscle torque when using a clinical electrical stimulator versus a portable electrical stimulator. Phys Ther. 2005 Jan;85(1):44-51. PMID 15623361
- [Background] Jaggers JR, Simpson CD, Frost KL, Quesada PM, Topp RV, Swank AM, Nyland JA. Prehabilitation before knee arthroplasty increases postsurgical function: a case study. J Strength Cond Res. 2007 May;21(2):632-4. doi: 10.1519/R-19465.1. PMID 17530958
- [Background] Svinoy OE, Bergland A, Risberg MA, Pripp AH, Hilde G. Better before-better after: efficacy of prehabilitation for older patients with osteoarthritis awaiting total hip replacement-a study protocol for a randomised controlled trial in South-Eastern Norway. BMJ Open. 2019 Dec 30;9(12):e031626. doi: 10.1136/bmjopen-2019-031626. PMID 31892650
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714